CLINICAL TRIAL: NCT03885791
Title: Randomized Controlled Trial of Vaginal Cryotherapy for Pelvic Floor Myofascial Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201901209
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Floor Myofascial Pain; Pelvic Pain; Myofascial Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal cryotherapy - intervention (Experimental): The intervention group will be provided with one vaginal cryotherapy tube, filled with a mixture of isopropyl alcohol (2ml) and water (8ml) that has been kept in the freezer. This mixture results in a "slushy" consistency and prevents the solution from freezing solid thus decreases the risk of discomfort or injury due to the temperature of the tube. Patients will insert this tube into the vagina to a comfortable depth. A lubricant will be provided for comfort with tube insertion, if necessary. At the conclusion of the treatment, this tube will be washed thoroughly and given to the patient in a clean plastic baggie for use at home. They will be instructed to store these tubes in their home freezer.
  Interventions: Device: vaginal cryotherapy
- Vaginal cryotherapy - control (Placebo Comparator): The control group will be provided with an identical tube that is empty. An empty tube was chosen as the control because a tube with room-temperature liquid may still be perceived as cold. Patients will insert this tube into the vagina to a comfortable depth. A lubricant will be provided for comfort with tube insertion, if necessary. At the conclusion of the treatment, this tube will be washed thoroughly and given to the patient in a clean plastic baggie for use at home. They will be instructed to store these tubes in their home at room temperature.
  Interventions: Device: vaginal cryotherapy

INTERVENTIONS:
Device: vaginal cryotherapy — Both groups will be given the same instructions for use, which will include intravaginal placement of one tube for 10 minutes while resting in a supine position. A lubricant may be used for comfort with insertion.
  Patients will perform their first intervention in the office with a repeat examination within 10 minutes of completing therapy. Patients participating in Specific Aims #2 will perform the intervention once daily at home. Patients will be asked to complete a short diary for each session, which will include the time of day, duration of application, pain score prior to and after application, and presence of any pelvic floor disorder symptoms prior to and after application.

SUMMARY:
This is a placebo-controlled, randomized controlled trial to investigate the role of vaginal cryotherapy on pelvic floor myofascial pain in women. This study involves randomizing patients who are found to have pelvic floor myofascial pain on examination into one of two treatment groups: transvaginal cryotherapy or transvaginal application of a room-temperature tube. Patients will be followed up at two different time points in order to assess response to treatment. Follow-up times include immediately after application (Specific Aim #1) and two weeks following use of the intervention alone (Specific Aim #2). Patients will receive verbal and written instructions on using the intravaginal tubes by the research assistant who will not be blinded to treatment allocation. Patients will not be blinded to their treatment assignment but will not be given information on the alternative treatment. Patients will be referred to pelvic floor PT, which is considered the standard of care for treatment of pelvic floor myofascial pain at this time. As it typically takes 2-3 weeks to get in to see one of the pelvic floor PT providers at Wash U, follow up for this study will be completed prior to their attendance at pelvic floor PT. Patients will complete validated questionnaires assessing their pain, other pelvic floor symptoms, and acceptance of the intervention as a treatment option at the follow up time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18yo)
* Women
* Patients found to have pelvic floor myofascial pain of at least 4/10 in severity at any of the four sites (right obturator internus, right levator ani, left levator ani, left obturator internus)

Exclusion Criteria:

* Age <18
* Non-English speaking
* Current diagnosis of dementia
* Limited physical mobility that would prevent full participation in pelvic floor PT.
* Prior use of vaginal cryotherapy
* Chief complaint or known history of pelvic pain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
change in myofascial pain score | 10-15 minutes (Pre- to post-treatment)
  Primary outcome is change in pelvic floor myofascial pain scores at each site (bilateral OI and LA) as measured on a 0-10 visual pain rating scale where 0 indicates no pain on palpation and 10 indicates 'worst pain imaginable' on palpation.

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory-20 | 2 weeks
  Short form of the validated questionnaire to assess presence and degree of bother of common pelvic floor symptoms
Pelvic Floor Impact Questionnaire-7 | 2 weeks
  Short form of the validated questionnaire to assess impact of pelvic floor symptoms on daily activities
Prolapse and Incontinence Sexual Questionnaire | 2 weeks
  Short form of the validated questionnaire to assess the impact of pelvic floor symptoms on sexual activity
Urogenital Distress Inventory | 2 weeks
  Validated questionnaire to assess presence and degree of bother of lower urinary tract symptoms
Lower Urinary Tract Symptoms (LUTS) Tool | 2 weeks
  Validated questionnaire to assess lower urinary tract symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Outpatient Health/Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sexton CC, Coyne KS, Kopp ZS, Irwin DE, Milsom I, Aiyer LP, Tubaro A, Chapple CR, Wein AJ; EpiLUTS Team. The overlap of storage, voiding and postmicturition symptoms and implications for treatment seeking in the USA, UK and Sweden: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:12-23. doi: 10.1111/j.1464-410X.2009.08369.x. PMID 19302498
- [Background] Adams K, Gregory WT, Osmundsen B, Clark A. Levator myalgia: why bother? Int Urogynecol J. 2013 Oct;24(10):1687-93. doi: 10.1007/s00192-013-2089-8. Epub 2013 Apr 11. PMID 23575699
- [Background] Pastore EA, Katzman WB. Recognizing myofascial pelvic pain in the female patient with chronic pelvic pain. J Obstet Gynecol Neonatal Nurs. 2012 Sep-Oct;41(5):680-91. doi: 10.1111/j.1552-6909.2012.01404.x. Epub 2012 Aug 3. PMID 22862153
- [Background] Spitznagle TM, Robinson CM. Myofascial pelvic pain. Obstet Gynecol Clin North Am. 2014 Sep;41(3):409-32. doi: 10.1016/j.ogc.2014.04.003. Epub 2014 Jul 9. PMID 25155122
- [Background] Borg-Stein J, Iaccarino MA. Myofascial pain syndrome treatments. Phys Med Rehabil Clin N Am. 2014 May;25(2):357-74. doi: 10.1016/j.pmr.2014.01.012. Epub 2014 Mar 17. PMID 24787338
- [Background] Bedaiwy MA, Patterson B, Mahajan S. Prevalence of myofascial chronic pelvic pain and the effectiveness of pelvic floor physical therapy. J Reprod Med. 2013 Nov-Dec;58(11-12):504-10. PMID 24568045
- [Background] Nadler SF, Weingand K, Kruse RJ. The physiologic basis and clinical applications of cryotherapy and thermotherapy for the pain practitioner. Pain Physician. 2004 Jul;7(3):395-9. PMID 16858479
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Kalder M, Pantazis K, Dinas K, Albert US, Heilmaier C, Kostev K. Discontinuation of treatment using anticholinergic medications in patients with urinary incontinence. Obstet Gynecol. 2014 Oct;124(4):794-800. doi: 10.1097/AOG.0000000000000468. PMID 25198276
- [Background] Latthe P, Latthe M, Say L, Gulmezoglu M, Khan KS. WHO systematic review of prevalence of chronic pelvic pain: a neglected reproductive health morbidity. BMC Public Health. 2006 Jul 6;6:177. doi: 10.1186/1471-2458-6-177. PMID 16824213
- [Background] Sedighimehr N, Manshadi FD, Shokouhi N, Baghban AA. Pelvic musculoskeletal dysfunctions in women with and without chronic pelvic pain. J Bodyw Mov Ther. 2018 Jan;22(1):92-96. doi: 10.1016/j.jbmt.2017.05.001. Epub 2017 May 3. PMID 29332764
- [Background] Peters KM, Carrico DJ. Frequency, urgency, and pelvic pain: treating the pelvic floor versus the epithelium. Curr Urol Rep. 2006 Nov;7(6):450-5. doi: 10.1007/s11934-006-0053-6. PMID 17052440
- [Background] Moldwin RM, Fariello JY. Myofascial trigger points of the pelvic floor: associations with urological pain syndromes and treatment strategies including injection therapy. Curr Urol Rep. 2013 Oct;14(5):409-17. doi: 10.1007/s11934-013-0360-7. PMID 23943509
- [Background] Biurrun Manresa JA, Neziri AY, Curatolo M, Arendt-Nielsen L, Andersen OK. Reflex receptive fields are enlarged in patients with musculoskeletal low back and neck pain. Pain. 2013 Aug;154(8):1318-24. doi: 10.1016/j.pain.2013.04.013. Epub 2013 Apr 9. PMID 23707309
- [Background] FitzGerald MP, Kotarinos R. Rehabilitation of the short pelvic floor. I: Background and patient evaluation. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Oct;14(4):261-8. doi: 10.1007/s00192-003-1049-0. Epub 2003 Aug 2. PMID 14530839
- [Background] White GE, Wells GD. Cold-water immersion and other forms of cryotherapy: physiological changes potentially affecting recovery from high-intensity exercise. Extrem Physiol Med. 2013 Sep 1;2(1):26. doi: 10.1186/2046-7648-2-26. PMID 24004719
- [Background] Ferreira-Junior JB, Bottaro M, Vieira A, Siqueira AF, Vieira CA, Durigan JL, Cadore EL, Coelho LG, Simoes HG, Bemben MG. One session of partial-body cryotherapy (-110 degrees C) improves muscle damage recovery. Scand J Med Sci Sports. 2015 Oct;25(5):e524-30. doi: 10.1111/sms.12353. Epub 2014 Dec 30. PMID 25556301
- [Background] Hohenauer E, Taeymans J, Baeyens JP, Clarys P, Clijsen R. The Effect of Post-Exercise Cryotherapy on Recovery Characteristics: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 28;10(9):e0139028. doi: 10.1371/journal.pone.0139028. eCollection 2015. PMID 26413718
- [Background] Rogers RG, Rockwood TH, Constantine ML, Thakar R, Kammerer-Doak DN, Pauls RN, Parekh M, Ridgeway B, Jha S, Pitkin J, Reid F, Sutherland SE, Lukacz ES, Domoney C, Sand P, Davila GW, Espuna Pons ME. A new measure of sexual function in women with pelvic floor disorders (PFD): the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1091-103. doi: 10.1007/s00192-012-2020-8. Epub 2013 Apr 30. PMID 23632798
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Rockwood TH, Constantine ML, Adegoke O, Rogers RG, McDermott E, Davila GW, Domoney C, Jha S, Kammerer-Doak D, Lukacz ES, Parekh M, Pauls R, Pitkin J, Reid F, Ridgeway B, Thakar R, Sand PK, Sutherland SE, Espuna-Pons M. The PISQ-IR: considerations in scale scoring and development. Int Urogynecol J. 2013 Jul;24(7):1105-22. doi: 10.1007/s00192-012-2037-z. Epub 2013 Apr 30. PMID 23632799
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Meister MR, Shivakumar N, Sutcliffe S, Spitznagle T, Lowder JL. Physical examination techniques for the assessment of pelvic floor myofascial pain: a systematic review. Am J Obstet Gynecol. 2018 Nov;219(5):497.e1-497.e13. doi: 10.1016/j.ajog.2018.06.014. Epub 2018 Jun 28. PMID 29959930
- [Background] Sutcliffe S, Bradley CS, Clemens JQ, James AS, Konkle KS, Kreder KJ, Lai HH, Mackey SC, Ashe-McNalley CP, Rodriguez LV, Barrell E, Hou X, Robinson NA, Mullins C, Berry SH. Urological chronic pelvic pain syndrome flares and their impact: qualitative analysis in the MAPP network. Int Urogynecol J. 2015 Jul;26(7):1047-60. doi: 10.1007/s00192-015-2652-6. Epub 2015 Mar 20. PMID 25792349
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03885791/Prot_SAP_000.pdf